CLINICAL TRIAL: NCT02252042
Title: A Phase III Randomized Trial of MK-3475 (Pembrolizumab) Versus Standard Treatment in Subjects With Recurrent or Metastatic Head and Neck Cancer
Brief Title: Pembrolizumab (MK-3475) Versus Standard Treatment for Recurrent or Metastatic Head and Neck Cancer (MK-3475-040/KEYNOTE-040)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-040; MK-3475-040 (Other: Merck Protocol Number); 2014-001749-26 (EudraCT Number)
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Cancer
Keywords: Squamous cell carcinoma; Head and neck carcinoma; Programmed Cell Death-1 (PD1, PD-1),; Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death Receptor Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Carcinoma, Squamous Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Methotrexate; Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembroliziumab (Experimental): Participants will receive pembrolizumab 200 mg intravenous (IV) on Day 1 of each 3-week cycle for up to approximately 24 months. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to approximately 1 additional year at the investigator's discretion.
  Interventions: Biological: Pembrolizumab
- Standard Treatment (Active Comparator): Participants will receive standard treatment of either methotrexate 40 mg/m^2 IV (may be escalated to 60 mg/m^2 maximum dose) on Days 1, 8, and 15 of each 3-week cycle; or docetaxel 75 mg/m^2 IV on Day 1 of each 3- week cycle; or cetuximab 400 mg/m^2 IV loading dose on Day 1 and 250 mg/m^2 IV on Days 8 and 15 of Cycle 1, followed by cetuximab 250 mg/m^2 on Days 1, 8, and 15 of each subsequent 3-week cycle.
  Interventions: Drug: Methotrexate; Drug: Docetaxel; Biological: Cetuximab

INTERVENTIONS:
Biological: Pembrolizumab — 200 mg intravenous (IV) on Day 1 of each 3-week cycle.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembroliziumab
Drug: Methotrexate — 40 mg/m^2 IV (may be escalated to 60 mg/m^2 maximum dose) on Days 1, 8, and 15 of each 3-week cycle
  Arms: Standard Treatment
Drug: Docetaxel — 75 mg/m^2 IV on Day 1 of each 3- week cycle
  Arms: Standard Treatment
Biological: Cetuximab — 400 mg/m^2 IV loading dose on Day 1 and 250 mg/m^2 IV on Days 8 and 15 of Cycle 1, followed by 250 mg/m^2 on Days 1, 8, and 15 of each subsequent 3-week cycle.
  Arms: Standard Treatment

SUMMARY:
This is a study of pembrolizumab (MK-3475, KEYTRUDA®) versus standard treatment (methotrexate, docetaxel or cetuximab) for the treatment of recurrent or metastatic head and neck squamous cell cancer (HNSCC). Participants will be randomly assigned to receive either pembrolizumab or Investigator's choice of standard treatment. The primary study hypothesis is that pembrolizumab treatment prolongs Overall Survival (OS) when compared to standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed recurrent disease not amenable to curative treatment with local or systemic therapy, or metastatic (disseminated) head and neck squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies
* Failure of prior platinum therapy
* Radiographically-measurable disease based on RECIST 1.1
* Tumor tissue available for PD-L1 biomarker analysis
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Female participants of childbearing potential must be willing to use 2 methods of birth control or abstain from heterosexual activity for the course of the study through 120 days after last dose of pembrolizumab or through 120-180 days after the last dose of docetaxel, methotrexate or cetuximab, acccording to local standard of care
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after last dose of pembrolizumab or through 120-180 days after the last dose of docetaxel, methotrexate or cetuximab, acccording to local standard of care

Exclusion Criteria

* Disease is suitable for local therapy administered with curative intent
* Currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks prior to randomization
* Previously treated with 3 or more systemic regimens given for recurrent and/or metastatic disease
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study therapy
* Not recovered from adverse events due to therapy more than 4 weeks earlier
* Prior anti-cancer monoclonal antibody (mAb) therapy within 4 weeks prior to study Day 1, or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1
* Diagnosed and/or treated additional malignancy within 5 years of randomization, with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, and/or curatively-resected in situ cervical and/or breast cancers
* Active autoimmune disease that has required systemic therapy in the past 2 years with modifying agents, corticosteroids, or immunosuppressive agents
* Active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial therapy according to local standard of care
* Prior therapy with an anti-PD-1 or anti-PD1-L1 or -L2 therapy or previously participated in a Merck pembrolizumab (MK-3475) trial
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* Live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2022-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Xin W, Ding H, Fang Q, Zheng X, Tong Y, Xu G, Yang G. Cost-effectiveness of pembrolizumab for treatment of platinum-resistant recurrent or metastatic head and neck squamous cell carcinoma in China: an economic analysis based on a randomised, open-label, phase III trial. BMJ Open. 2020 Dec 18;10(12):e038867. doi: 10.1136/bmjopen-2020-038867. PMID 33371020
- [Derived] Emancipator K, Huang L, Aurora-Garg D, Bal T, Cohen EEW, Harrington K, Soulieres D, Le Tourneau C, Licitra L, Burtness B, Swaby R. Comparing programmed death ligand 1 scores for predicting pembrolizumab efficacy in head and neck cancer. Mod Pathol. 2021 Mar;34(3):532-541. doi: 10.1038/s41379-020-00710-9. Epub 2020 Nov 25. PMID 33239737
- [Derived] Pai SI, Faivre S, Licitra L, Machiels JP, Vermorken JB, Bruzzi P, Gruenwald V, Giglio RE, Leemans CR, Seiwert TY, Soulieres D. Comparative analysis of the phase III clinical trials of anti-PD1 monotherapy in head and neck squamous cell carcinoma patients (CheckMate 141 and KEYNOTE 040). J Immunother Cancer. 2019 Apr 3;7(1):96. doi: 10.1186/s40425-019-0578-0. PMID 30944020
- [Derived] Cohen EEW, Soulieres D, Le Tourneau C, Dinis J, Licitra L, Ahn MJ, Soria A, Machiels JP, Mach N, Mehra R, Burtness B, Zhang P, Cheng J, Swaby RF, Harrington KJ; KEYNOTE-040 investigators. Pembrolizumab versus methotrexate, docetaxel, or cetuximab for recurrent or metastatic head-and-neck squamous cell carcinoma (KEYNOTE-040): a randomised, open-label, phase 3 study. Lancet. 2019 Jan 12;393(10167):156-167. doi: 10.1016/S0140-6736(18)31999-8. Epub 2018 Nov 30. PMID 30509740
- [Derived] Guo T, Califano JA. Molecular biology and immunology of head and neck cancer. Surg Oncol Clin N Am. 2015 Jul;24(3):397-407. doi: 10.1016/j.soc.2015.03.002. Epub 2015 Apr 20. PMID 25979390
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 495 participants were randomized 1:1 to receive either pembrolizumab or standard treatment. Per protocol, response/progression or adverse events (AEs) that occurred during the second course of pembrolizumab were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg intravenous (IV) on Day 1 of each 3-week cycle. Eligible participants who stopped the initial course of pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Standard Treatment: Participants received standard treatment of either methotrexate 40 mg/m^2 IV (could be escalated to 60 mg/m^2 maximum dose) on Days 1, 8, and 15 of each 3-week cycle; or docetaxel 75 mg/m^2 IV on Day 1 of each 3- week cycle; or cetuximab 400 mg/m^2 IV loading dose on Day 1 and 250 mg/m^2 IV on Days 8 and 15 of Cycle 1, followed by cetuximab 250 mg/m^2 on Days 1, 8, and 15 of each subsequent 3-week cycle.
Period: Overall Study
Arm/Group | Pembrolizumab | Standard Treatment
Started | 247 | 248
Received First Course of Pembrolizumab | 246 (1 participant was randomized but did not receive study treatment.) | 234 (14 participants were randomized but did not receive study treatment.)
Received Second Course of Pembrolizumab | 2 | 0
Completed | 0 | 0
Not Completed | 247 | 248
Not completed — Adverse Event | 9 | 6
Not completed — Death | 209 | 217
Not completed — Physician Decision | 0 | 2
Not completed — Transferred to Extension Study | 7 | 1
Not completed — Did Not Continue on Extension Study | 7 | 2
Not completed — Withdrawal by Subject | 15 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab | Standard Treatment | Total
Number analyzed (Participants) | 247 | 248 | 495
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (9.8) | 60.2 (8.6) | 60.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 207 | 205 | 412
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 12 | 33
  Not Hispanic or Latino | 182 | 195 | 377
  Unknown or Not Reported | 44 | 41 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants] — The race of participants is presented.
  Participants
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 15 | 16 | 31
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 7 | 10
    White | 206 | 207 | 413
    More than one race | 4 | 3 | 7
    Unknown or Not Reported | 17 | 15 | 32
Programmed Cell Death-Ligand 1 (PD-L1) Expression Level: Tumor Proportion Score (TPS) [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a TPS ≥50% were classified as PD-L1 strongly positive and participants with a TPS <50% were classified as not strongly positive.
  Participants
    TPS = 0% | 103 | 93 | 196
    1% ≤ TPS <50% | 79 | 87 | 166
    TPS ≥ 50% | 64 | 65 | 129
    Missing | 1 | 3 | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were assessed for ECOG PS: Grade 0: Fully active, able to carry on all pre-disease performance without restriction; Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light or sedentary nature; Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities, up & about more than 50% of waking hours; Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; Grade 4: Completely disabled, cannot carry on any selfcare, totally confined to bed or chair or Grade 5: Dead.
  Participants
    EGOG PS=0 | 71 | 68 | 139
    ECOG PS=1 | 176 | 179 | 355
    ECOG PS=2 | 0 | 1 | 1
Human Papillomavirus (HPV) Tumor Status [Count of Participants; unit: Participants] — Participants were assessed for the presence or absence of HPV in their tumors.
  Participants
    Positive HPV Status | 61 | 57 | 118
    Negative HPV Status | 186 | 191 | 377
PD-L1 Combined Positive Score (CPS) Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from a newly obtained biopsy. Participants with a CPS ≥1 were classified as PD-L1 positive and participants with a CPS <1 were classified as PD-L1 negative.
  Participants
    PD-L1 CPS <1 | 50 | 54 | 104
    PD-L1 CPS ≥1 | 196 | 191 | 387
    Missing | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Initial Overall Survival (OS) for All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The OS for all participants is presented. These initial OS results are based on a data cutoff date of 15-May-2017 with a database lock date of 04-Jun-2017. At the time of the database lock of 04-Jun-2017, there was incomplete collection of survival data for 12 participants.
Time Frame: Up to approximately 2 years
Population: The efficacy population consisted of all randomized participants. Participants are included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Months | 8.4 [6.5 to 9.4] | 7.1 [5.9 to 8.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.03160, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.67 to 1.01] — Cox regression model with treatment as a covariate stratified by ECOG PS (0 vs. 1), HPV status (Positive vs. Negative) & PD-L1 status (Strongly Positive, Not Strongly Positive)

2. Primary Outcome: Updated Final OS for All Participants
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were to be censored at the date of the last follow-up. The updated OS for all participants is presented. These OS results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Months | 8.4 [6.4 to 9.4] | 6.9 [5.9 to 8.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.01605, Log Rank — Nominal p-value; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.65 to 0.98] — Nominal HR. Cox regression model with treatment as a covariate stratified by ECOG PS (0 vs. 1), HPV status (Positive vs. Negative) & PD-L1 status (Strongly Positive, Not Strongly Positive)

3. Secondary Outcome: OS for Participants With Programmed Cell Death-Ligand 1 (PD-L1)-Positive Expression Defined by ≥1% Combined Positive Score (CPS)(PD-L1 ≥1% CPS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. The OS for all participants with PD-L1 expression ≥1% CPS was presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: The efficacy population consisted of all randomized participants with PD-L1 ≥1% CPS. Participants are included in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 196 | 191
Months | 8.7 [6.9 to 11.4] | 7.1 [5.7 to 8.3]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.00493, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.58 to 0.93] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 for All Participants
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded central imaging vendor review or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. The PFS per RECIST 1.1 for all participants is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Months | 2.1 [2.1 to 2.3] | 2.3 [2.1 to 2.8]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.32504, Log Rank; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.79 to 1.16] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: PFS Per RECIST 1.1 in Participants With PD-L1 ≥1% CPS
Description: PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded central imaging vendor review or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. The PFS per RECIST 1.1 for all participants with PD-L1 expression ≥1% CPS is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 196 | 191
Months | 2.2 [2.1 to 3.0] | 2.3 [2.1 to 3.0]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.07736, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.69 to 1.06] — Cox regression model with treatment as a single covariate

6. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1 in All Participants
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based on blinded central imaging vendor review with or without confirmation. The ORR per RECIST 1.1 for all participants is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Percentage of Participants | 14.6 [10.4 to 19.6] | 10.1 [6.6 to 14.5]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.0610, Log Rank; H0: difference in %=0; H1: difference in %>0; Difference in percentages = 4.6, 95% CI 2-sided [-1.2 to 10.6] — Stratified by ECOG PS (0 vs. 1), HPV status (Positive vs. Negative) & PD-L1 status (Strongly Positive, Not Strongly Positive)

7. Secondary Outcome: ORR Per RECIST 1.1 in Participants With PD-L1 ≥1% CPS
Description: ORR was defined as the percentage of the participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1 based on blinded central imaging vendor review with or without confirmation. The ORR per RECIST 1.1 for all participants with PD-L1 expression ≥1% CPS is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 196 | 191
Percentage of Participants | 17.3 [12.3 to 23.4] | 9.9 [6.1 to 15.1]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.0171, Log Rank; H0: difference in %=0; H1: difference in %>0; Difference in percentages = 7.5, 95% CI 2-sided [0.6 to 14.6] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 in All Participants
Description: For participants who demonstrated a confirmed CR or PR per RECIST 1.1, DOR was defined as the time from first documented evidence of a confirmed CR or PR per RECIST 1.1 until disease progression per RECIST 1.1 or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. DOR assessments were based on blinded central imaging vendor review with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: The efficacy population consisted of all randomized participants who demonstrated a confirmed CR or PR per RECIST 1.1. Participants are included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 26 | 18
Months | 18.4 [2.7 to 18.4] | 5.0 [1.4 to 18.8]

9. Secondary Outcome: DOR Per RECIST 1.1 in Participants With PD-L1 ≥1% CPS
Description: For participants who demonstrated a confirmed CR or PR per RECIST 1.1, DOR was defined as the time from first documented evidence of a confirmed CR or PR per RECIST 1.1 until disease progression per RECIST 1.1 or death due to any cause, whichever occurred first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. DOR assessments were based on blinded central imaging vendor review with confirmation. The DOR per RECIST 1.1 for all participants with PD-L1 ≥1% CPS who experienced a confirmed CR or PR is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: The efficacy population consisted of all randomized participants with PD-L1 ≥1% CPS who demonstrated a confirmed CR or PR per RECIST 1.1. Participants are included in the treatment group to which they were randomized.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 26 | 15
Months | 18.4 [2.7 to 18.4] | 9.6 [1.4 to 18.8]

10. Secondary Outcome: Time to Progression (TTP) Per RECIST 1.1 in All Participants
Description: TTP was defined as the time from randomization to the first documented disease progression based on assessments by the blinded central imaging vendor review per RECIST 1.1. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. The TTP per RECIST 1.1 for all participants is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Months | 2.2 [2.1 to 3.3] | 2.2 [2.1 to 3.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.14545, Log Rank — p-value stratified by ECOG PS (0 vs. 1), HPV status (Positive vs. Negative) & PD-L1 status (Strongly Positive, Not Strongly Positive); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.70 to 1.12] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: TTP Per RECIST 1.1 in Participants With PD-L1 ≥1% CPS
Description: TTP was defined as the time from randomization to the first documented disease progression based on assessments by the blinded central imaging vendor review per RECIST 1.1. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. The TTP per RECIST 1.1 for all participants with PD-L1 ≥1% CPS is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 196 | 191
Months | 2.7 [2.1 to 3.5] | 2.3 [2.1 to 3.4]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.05851, Log Rank — [p-value comment as in outcome 10, analysis 1]; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.62 to 1.06] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: PFS Per Modified RECIST in All Participants
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on blinded central imaging vendor review or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. Modified RECIST is similar to RECIST 1.1 with the exception that a confirmation assessment of PD (>4 weeks after the initial PD) is required for participants who remain on treatment following a documented PD per RECIST 1.1. The PFS per modified RECIST for all participants is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 247 | 248
Months | 3.5 [3.1 to 4.4] | 4.8 [4.1 to 5.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.65759, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.86 to 1.27] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: PFS Per Modified RECIST 1.1 in Participants With PD-L1 ≥1% CPS
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on blinded central imaging vendor review or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. Modified RECIST is similar to RECIST 1.1 with the exception that a confirmation assessment of PD (>4 weeks after the initial PD) is required for participants who remain on treatment following a documented PD per RECIST 1.1. The PFS per modified RECIST for all participants with PD-L1 ≥1% CPS is presented. These efficacy results were reported after complete acquisition of all outstanding survival data using a 15-May-2017 data cut-off date with a database update date of 13-Oct-2017.
Time Frame: Up to approximately 2 years
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 196 | 191
Months | 3.6 [3.1 to 4.6] | 4.8 [4.1 to 5.7]
Statistical Analysis 1: Comparison: Pembrolizumab vs Standard Treatment; Test type: Superiority; p = 0.51982, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.81 to 1.26] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Number of Participants Who Experienced At Least One Adverse Event (AE) in All Participants
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants who experienced at least one AE is presented.
Time Frame: Up to approximately 33 months
Population: The safety population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 246 | 234
Participants | 240 | 227

15. Secondary Outcome: Number of Participants Who Experienced At Least One AE in Participants With PD-L1 ≥1% CPS
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants with PD-L1 ≥1% CPS who experienced at least one AE is presented.
Time Frame: Up to approximately 33 months
Population: The safety population consisted of all randomized participants with PD-L1 ≥1% CPS who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 195 | 183
Participants | 193 | 178

16. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE in All Participants
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 30 months
Population: The safety population consisted of all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 246 | 234
Participants | 30 | 36

17. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE in Participants With PD-L1 ≥1% CPS
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE. The number of all participants with PD-L1 ≥1% CPS who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 30 months
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab | Standard Treatment
Number analyzed (Participants) | 195 | 183
Participants | 25 | 29

ADVERSE EVENTS:
Time Frame: Up to approximately 92 months
Description: All-Cause Mortality was reported for all randomized participants.
  Serious AEs and Other AEs were reported according to treatment course for all randomized participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer on study was not considered an AE unless considered related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Pembrolizumab First Course: Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for up to approximately 24 months.
- Standard Treatment First Course: Participants received standard treatment of either methotrexate 40 mg/m^2 IV (could be escalated to 60 mg/m^2 maximum dose) on Days 1, 8, and 15 of each 3-week cycle; or docetaxel 75 mg/m^2 IV on Day 1 of each 3- week cycle; or cetuximab 400 mg/m^2 IV loading dose on Day 1 and 250 mg/m^2 IV on Days 8 and 15 of Cycle 1, followed by cetuximab 250 mg/m^2 on Days 1, 8, and 15 of each subsequent 3-week cycle.
- Pembrolizumab Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to approximately 24 months) with SD or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to approximately 1 additional year.
Arm/Group | Pembrolizumab First Course | Standard Treatment First Course | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 228/247 | 243/248 | 2/2
Serious Adverse Events (participants affected / at risk) | 110/246 | 92/234 | 0/2
Other Adverse Events (participants affected / at risk) | 215/246 | 211/234 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=246) | Standard Treatment First Course (N=234) | Pembrolizumab Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 0 (0)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 9 (9) | 0 (0)
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 3 (3) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (7) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 4 (4) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral discharge (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 5 (5) | 4 (4) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 3 (3) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 22 (23) | 17 (19) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 6 (7) | 3 (3) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Stoma site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Stoma site ulcer (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheostomy malfunction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 3 (5) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Soft tissue haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10) | 2 (4) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0)
Eosinophilic pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fungating wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Euthanasia (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Angiodysplasia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab First Course (N=246) | Standard Treatment First Course (N=234) | Pembrolizumab Second Course (N=2)
Anaemia (Blood and lymphatic system disorders) | 61 (77) | 53 (72) | 0 (0)
Hypothyroidism (Endocrine disorders) | 41 (45) | 10 (10) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (12) | 12 (12) | 0 (0)
Constipation (Gastrointestinal disorders) | 43 (49) | 37 (43) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 37 (57) | 42 (51) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 15 (15) | 6 (6) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 21 (22) | 15 (16) | 0 (0)
Nausea (Gastrointestinal disorders) | 36 (45) | 44 (52) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 7 (9) | 26 (34) | 0 (0)
Vomiting (Gastrointestinal disorders) | 24 (28) | 23 (34) | 0 (0)
Asthenia (General disorders) | 40 (50) | 42 (54) | 0 (0)
Fatigue (General disorders) | 49 (53) | 63 (81) | 0 (0)
Mucosal inflammation (General disorders) | 17 (21) | 36 (51) | 0 (0)
Pyrexia (General disorders) | 24 (38) | 25 (36) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (10) | 13 (18) | 0 (0)
Lymphocyte count decreased (Investigations) | 13 (16) | 10 (13) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (11) | 24 (29) | 0 (0)
Platelet count decreased (Investigations) | 7 (7) | 13 (19) | 0 (0)
Weight decreased (Investigations) | 21 (24) | 25 (25) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 31 (37) | 45 (50) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 14 (16) | 13 (14) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 23 (27) | 19 (21) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 10 (11) | 20 (25) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (14) | 16 (17) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 15 (21) | 12 (14) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (24) | 12 (13) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (24) | 8 (8) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 20 (20) | 17 (17) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 7 (8) | 0 (0)
Headache (Nervous system disorders) | 21 (25) | 23 (25) | 0 (0)
Anxiety (Psychiatric disorders) | 13 (13) | 7 (7) | 0 (0)
Insomnia (Psychiatric disorders) | 22 (22) | 18 (18) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (49) | 37 (40) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 (33) | 26 (31) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 7 (9) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 5 (7) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 27 (27) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 18 (28) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4) | 17 (19) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (24) | 17 (40) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 26 (33) | 41 (92) | 0 (0)
Hypotension (Vascular disorders) | 13 (13) | 12 (16) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT02252042/Prot_SAP_001.pdf